CLINICAL TRIAL: NCT04900363
Title: A Phase Ib/II Trial of AK112 (PD-1/VEGF Bispecific Antibody) in Patients With Advanced NSCLC
Brief Title: A Trial of AK112 (PD-1/VEGF Bispecific Antibody) in Patients With NSCLC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-202
Record Dates: First submitted 2021-04-29; First posted 2021-05-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK112 (Experimental): Subjects receive AK112 monotherapy intravenously (IV) until no more benefits from treatment.
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — Subjects receive AK112 intravenously.

SUMMARY:
This trial is a Phase Ib/II study. All patients are stage IIIB/C or IV non-small cell lung cancer(NSCLC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of AK112 in subjects with advanced NSCLC whose tumors have a programmed cell death-ligand 1 (PD-L1) Tumor Proportion Score (TPS) greater than or equal to 1%.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of NSCLC.
* Has StageIIIB/C or IV NSCLC (American Joint Committee on Cancer [AJCC]).
* 18 to 75 years old (at the time consent is obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy.
* Has a life expectancy of at least 3 months.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team.
* Has adequate organ function.
* Has recovered from the effects of any prior radiotherapy or surgery.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Is currently participating in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment.
* Has undergone major surgery within 30 days of Study Day 1.
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases.
* Has carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to day 1 of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.
Number of participants with adverse events (AEs) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1
Duration of response (DOR) | up to 2 years
  Duration of response (DOR) assessed according to RECIST v1.1
Overall survival (OS) | up to 2 years
  Overall survival is defined as the time from the start of treatment with AK112 until death due to any cause.
Maximum observed concentration (Cmax) of AK112 | Up to 2 years
  Serum concentrations of AK112 in individual subjects at different time points after AK112 administration
Anti-drug antibodies (ADA) | Up to 2 years
  Number of subjects with detectable anti-drug antibodies (ADA)
PD-L1 expression | Up to 2 years
  The correlationship between PD-L1 expression and AK112 anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang L, Luo Y, Ren S, Zhang Z, Xiong A, Su C, Zhou J, Yu X, Hu Y, Zhang X, Dong X, Meng S, Wu F, Hou X, Dai Y, Song W, Li B, Wang ZM, Xia Y, Zhou C. A Phase 1b Study of Ivonescimab, a Programmed Cell Death Protein-1 and Vascular Endothelial Growth Factor Bispecific Antibody, as First- or Second-Line Therapy for Advanced or Metastatic Immunotherapy-Naive NSCLC. J Thorac Oncol. 2024 Mar;19(3):465-475. doi: 10.1016/j.jtho.2023.10.014. Epub 2023 Oct 23. PMID 37879536